CLINICAL TRIAL: NCT01727440
Title: Identifying the Genetic Predictors of Severe Acne Vulgaris and the Outcome of Oral Isotretinoin Treatment
Acronym: SA
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00030862
Record Dates: First submitted 2012-10-24; First posted 2012-11-16 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-01

CONDITIONS: Acne Vulgaris; Isotretinoin
Keywords: severe acne; severe acne vulgaris; acne; acne vulgaris; isotretinoin; Accutane; Sortret; Amnesteem; Claravis; Clarus; Decutan; Isotane; Izotek; Oratane; Isotret; Roaccutane
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood collected in three 2-mL EDTA tubes
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to enroll 250 participants that have joined the MURDOCK Study Horizon 1.5 (Duke IRB Pro00011196) with a current or prior diagnosis of severe acne AND current or prior treatment with oral isotretinoin. All 250 participants will answer a 5-page questionnaire designed to collect information on the diagnosis of severe acne and response to oral isotretinoin treatment. The aim is to identify genetic predictors of severe acne vulgaris and the outcome of oral isotretinoin treatment.

DETAILED DESCRIPTION:
Acne vulgaris is an under-studied common genetic disease with tremendous economic consequences. Acne vulgaris is one of the most common skin conditions treated by doctors. It affects 40-50 million people in the USA, with prevalence as high as 85% (recent study from Iran was 93%) in teenagers; 18% of woman have late onset (>25yr) acne vulgaris. Severe acne has a life-long psychosocial impact due to the significant scarring. Severe acne can also be associated with severe systemic inflammatory disease with fever, sterile osteomyelitis, inflammatory arthritis and other signs of systemic inflammatory responses. Some of these syndromes in Mendelian form (e.g. PAPA syndrome) have known genetic defects. Finally, while the data are inconclusive, there have been many suggestions that diet can exacerbate acne in some patients. The standard of care treatment for severe acne is systemic retinoid therapy, which, is usually, but not always effective. Unfortunately, systemic retinoid treatment is associated with significant toxicity, including common cutaneous adverse effects (dry lips, eyes, skin fragility), less common laboratory abnormalities such as elevated blood lipids, liver function abnormalities, and severe predictable teratogenicity. In addition, systemic therapy with retinoids has been associated with systemic diseases such as clinical depression, suicide, and inflammatory bowel disease, however the mechanisms and significance of these associations has not been determined. Given the frequency and severity of severe acne, the predictable severe toxicity of systemic retinoid therapy, and the already demonstrated genetic associations found in Mendelian forms of severe acne, it seems likely that significant genetic risk factors may be identified in patients with severe acne which would promote new and safer therapy, including dietary adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe acne while age > 12 and < 18, and
* Completed at least one course of oral isotretinoin treatment; OR started treatment but discontinued prior to completion due to adverse side effects (with the exception of dry skin - see "exclusion criteria"); OR are currently undergoing and plan to complete treatment

Exclusion Criteria:

* Patients who are not willing to participate in this study
* Patients who experienced inflammatory bowel disease (IBD) prior to oral isotretinoin treatment
* Patients who did not complete the oral isotretinoin treatment because of pregnancy, dry skin, or reasons other than adverse side effects listed above
* Patients who are not willing to or cannot provide a blood sample for Murdock Study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants must enroll or have enrolled in the MURDOCK Study Community Registry and Biorepository prior to joining this Severe Acne Study. At the MURDOCK Study visit, or after the participant has enrolled in the MURDOCK Study, they will be asked (either in person or via phone) if they would be willing to join the Severe Acne Study.
  Participants between ages 12 and 18 may also join the MURDOCK Study if they meet the eligibility criteria for this Severe Acne Study (a pediatric consent form will be used).
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Therapeutic response to isotretinoin | 10 months
  All 250 patients with severe acne will be genotyped using the Illumina 610 BeadChip. Whole-exome sequencing will be performed on 100 extremely severe acne vulgaris patients, selected based on severity and response to oral isotretinoin treatment. A case-control GWAS analysis will be performed (250 recruited patients vs. 1000 normal controls of convenience available in other studies at CHGV). Additionally, an association analyses will be conducted using complete exome sequencing data for the most severe cases, compared with controls of convenience (as an extreme trait in the population, there is a reasonable expectation of discovery of any important variants, rare or common). This analysis would also include targeted analysis on available drug response data (efficacy and adverse response).

SECONDARY OUTCOMES:
Adverse reaccion to isotretinoin | 10 months
  All 250 patients with severe acne will be genotyped using the Illumina 610 BeadChip. Whole-exome sequencing will be performed on 100 extremely severe acne vulgaris patients, selected based on severity and response to oral isotretinoin treatment. A case-control GWAS analysis will be performed (250 recruited patients vs. 1000 normal controls of convenience available in other studies at CHGV). Additionally, an association analyses will be conducted using complete exome sequencing data for the most severe cases, compared with controls of convenience (as an extreme trait in the population, there is a reasonable expectation of discovery of any important variants, rare or common). This analysis would also include targeted analysis on available drug response data (efficacy and adverse response).

CONTACTS AND LOCATIONS:
Overall Officials: Russell Hall, MD, Principal Investigator — Duke Medicine Site Based Research Group
Locations (6):
- United States (6):
  - Carolinas Medical Center Northeast Medical Arts Building, Concord, North Carolina
  - Dermatology Group of the Carolinas, Concord, North Carolina
  - Ada Jenkins Center, Davidson, North Carolina
  - Harrisburg Sleep Center, Harrisburg, North Carolina
  - Lake Norman Community Health Clinic, Huntersville, North Carolina
  - Kannapolis Internal Medicine, Kannapolis, North Carolina

REFERENCES:
- See also: Murdock Study Severe Acne Study — http://www.murdock-study.com/new-studies/severe-acne